CLINICAL TRIAL: NCT03036124
Title: Study to Evaluate the Effect of Dapagliflozin on the Incidence of Worsening Heart Failure or Cardiovascular Death in Patients With Chronic Heart Failure With Reduced Ejection Fraction
Brief Title: Study to Evaluate the Effect of Dapagliflozin on the Incidence of Worsening Heart Failure or Cardiovascular Death in Patients With Chronic Heart Failure
Acronym: DAPA-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1699C00001; 2016-003897-41 (EudraCT Number)
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction (HFrEF)
Keywords: HFrEF; Heart Failure (HF); Cardiovascular Events (CV); Phase III outcome trial
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Patients will be randomized 1:1 to either dapagliflozin or placebo.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo matching dapagliflozin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg or 5 mg tablets given once daily, per oral use.
  Other Names: Forxiga TM; Farxiga TM
  Arms: Dapagliflozin
Drug: Placebo — Placebo matching dapagliflozin 10 mg or 5 mg.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of dapagliflozin on the incidence of worsening heart failure or cardiovascular death in patients with chronic heart failure with reduced ejection fraction

DETAILED DESCRIPTION:
This is an international, multicentre, parallel group, event-driven, randomized, double-blind, placebo-controlled study in patients with chronic heart failure with reduced ejection fraction (HFrEF), evaluating the effect of dapagliflozin versus placebo, given once daily in addition to background regional standard of care therapy, for the prevention of cardiovascular (CV) death or reduction of heart failure (HF) events.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent prior to any study specific procedures
* Male or female, aged ≥18 years
* Established documented diagnosis of symptomatic HFrEF (NYHA functional class II-IV), which has been present for at least 2 months
* LVEF≤40%
* Elevated NT-proBNP levels
* Patients should receive background standard of care for HFrEF and be treated according to locally recognized guidelines
* eGFR ≥30 mL/min/1.73 m^2 (CKD-EPI formula) at enrolment (visit 1)

Exclusion Criteria:

* Receiving therapy with an SGLT2 inhibitor within 8 weeks prior to enrolment or previous intolerance of an SGLT2 inhibitor
* Type 1 diabetes mellitus
* Symptomatic hypotension or systolic BP <95 mmHg at 2 out of 3 measurements either at visit 1 or visit 2
* Current acute decompensated HF or hospitalization due to decompensated HF <4 weeks prior to enrolment
* MI, unstable angina, stroke or transient ischemic attack within 12 weeks prior to enrolment
* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) or valvular repair/replacement within 12 weeks prior to enrolment or planned to undergo any of these operations after randomization
* Implantation of a CRT within 12 weeks prior to enrolment or intent to implant a CRT device
* Previous cardiac transplantation or implantation of a ventricular assistance device or similar device, or implantation expected after randomization
* HF due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy or uncorrected primary valvular disease
* Symptomatic bradycardia or second or third degree heart block without a pacemaker
* Severe (eGFR <30 mL/min/1.73 m^2 by CKD-EPI), unstable or rapidly progressing renal disease at the time of randomization

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4744 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (333):
- United States (77):
  - Research Site, Fairhope, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Bakersfield, California
  - Research Site, Beverly Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Palm Springs, California
  - Research Site, Stockton, California
  - Research Site, Torrance, California
  - Research Site, Vista, California
  - Research Site, Wilmington, Delaware
  - Research Site, Boynton Beach, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, New Smyrna Beach, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, Wellington, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Cumming, Georgia
  - Research Site, Tucker, Georgia
  - Research Site, Hazel Crest, Illinois
  - Research Site, Jerseyville, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Chalmette, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, Flint, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Bridgewater, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Somerset, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Cortlandt Manor, New York
  - Research Site, New York, New York
  - Research Site, Orchard Park, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Rosedale, New York
  - Research Site, The Bronx, New York
  - Research Site, Burlington, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Altoona, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Rapid City, South Dakota
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Beaumont, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Farmington, Utah
  - Research Site, Falls Church, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
- Argentina (19):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Caba
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Ciudad Autonoma de Buenos Aire
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Esperanza
  - Research Site, Mar del Plata
  - Research Site, Quilmes
  - Research Site, Ramos Mejía
  - Research Site, Rosario
  - Research Site, San Luis
  - Research Site, San Martín
  - Research Site, San Miguel de Tucumán
  - Research Site, San Nicolás
  - Research Site, Santa Fe
  - Research Site, Vicente López
- Brazil (14):
  - Research Site, Belo Horizonte
  - Research Site, Brasillia
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Marília
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Uberlândia
  - Research Site, Votuporanga
- Bulgaria (8):
  - Research Site, Blagoevgrad
  - Research Site, Dimitrovgrad
  - Research Site, Haskovo
  - Research Site, Kyustendil
  - Research Site, Lom
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (25):
  - Research Site, Calgary, Alberta
  - Research Site, Abbotsford, British Columbia
  - Research Site, New Westminster, British Columbia
  - Research Site, North Vancouver, British Columbia
  - Research Site, Moncton, New Brunswick
  - Research Site, Saint John, New Brunswick
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Port Perry, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, York, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Rimouski, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Terrebonne, Quebec
- China (22):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chifeng
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Haerbin
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Pingxiang
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xuzhou
  - Research Site, Yinchuan
  - Research Site, Zhuhai
- Czechia (8):
  - Research Site, Benešov
  - Research Site, Brno
  - Research Site, Kolín
  - Research Site, Louny
  - Research Site, Ostrava-Dubina
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Třebíč
- Denmark (6):
  - Research Site, Hellerup
  - Research Site, Herlev
  - Research Site, Hvidovre
  - Research Site, København Ø
  - Research Site, Odense C
  - Research Site, Svendborg
- Germany (11):
  - Research Site, Bad Oeynhausen
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Hamburg
  - Research Site, Homburg
  - Research Site, Kassel
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Papenburg
  - Research Site, Stuttgart
  - Research Site, Wermsdorf
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Kecskemét
  - Research Site, Mosonmagyaróvár
  - Research Site, Szentes
  - Research Site, Székesfehérvár
  - Research Site, Zalaegerszeg
- India (14):
  - Research Site, Ahmedabad
  - Research Site, Aurangabad
  - Research Site, Bangalore
  - Research Site, Belagavi
  - Research Site, Ernākulam
  - Research Site, Gūrgaon
  - Research Site, Kanpur
  - Research Site, Karamsad
  - Research Site, Kolkata
  - Research Site, Maharashtra
  - Research Site, Nadiād
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Pune
- Japan (57):
  - Research Site, Adachi-ku
  - Research Site, Aki-gun,
  - Research Site, Azumino-shi
  - Research Site, Beppu-shi
  - Research Site, Bunkyō City
  - Research Site, Chikushino-shi
  - Research Site, Chūōku
  - Research Site, Fujisawa-shi
  - Research Site, Fukuoka
  - Research Site, Hachioji-shi
  - Research Site, Hamamatsu
  - Research Site, Himeji-shi
  - Research Site, Hiratsuka-shi
  - Research Site, Hitachi-Naka
  - Research Site, Iizuka-shi
  - Research Site, Itabashi-ku
  - Research Site, Iwakuni-shi
  - Research Site, Kagoshima
  - Research Site, Kakamigahara-shi
  - Research Site, Kasama-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kitakyusyu-shi
  - Research Site, Kumamoto
  - Research Site, Kure-shi
  - Research Site, Kusatsu-shi
  - Research Site, Kyoto
  - Research Site, Matsudo-shi
  - Research Site, Matsumoto-shi
  - Research Site, Matsuyama
  - Research Site, Meguro-ku
  - Research Site, Mito
  - Research Site, Miura-gun
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Nishinomiya-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sagamihara-shi
  - Research Site, Sakai-shi,Kita-ku
  - Research Site, Sakaide-shi
  - Research Site, Sanyoonoda-shi
  - Research Site, Sayama-shi
  - Research Site, Sendai
  - Research Site, Shimonoseki-shi
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Suwa-shi
  - Research Site, Tachikawa-shi
  - Research Site, Takamatsu
  - Research Site, Takasaki-shi
  - Research Site, Toride-shi
  - Research Site, Tsuchiura-shi
  - Research Site, Tsukuba
  - Research Site, Ueda-shi
  - Research Site, Wakayama
  - Research Site, Wako-shi
  - Research Site, Yokohama
- Netherlands (9):
  - Research Site, 's-Hertogenbosch
  - Research Site, Apeldoorn
  - Research Site, Gouda
  - Research Site, Groningen
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Sneek
  - Research Site, The Hague
  - Research Site, Veldhoven
- Poland (14):
  - Research Site, Bochnia
  - Research Site, Gdynia
  - Research Site, Jasło
  - Research Site, Katowice
  - Research Site, Kędzierzyn-Koźle
  - Research Site, Krakow
  - Research Site, Legnica
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Oława
  - Research Site, Płock
  - Research Site, Sokółka
  - Research Site, Torun
  - Research Site, Wierzchosławice
- Russia (10):
  - Research Site, Gatchina
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Perm
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Tver'
  - Research Site, Yekaterinburg
- Slovakia (10):
  - Research Site, Brezno
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Martin
  - Research Site, Nové Zámky
  - Research Site, Prešov
  - Research Site, Svidník
  - Research Site, Trebišov
  - Research Site, Trnava
  - Research Site, Žilina
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Östersund
  - Research Site, Stockholm
  - Research Site, Umeå
- Taiwan (7):
  - Research Site, Changhua
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Kweishan Shiang
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- United Kingdom (9):
  - Research Site, Airdrie
  - Research Site, Clydebank
  - Research Site, Cottingham
  - Research Site, Dundee
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Inverness
  - Research Site, Nottingham
  - Research Site, Paisley
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Myte R, Mattsson A, Poole M, Little DJ, Nystrom P, Henderson A, Claggett BL, Gasparyan SB, Solomon SD, McMurray JJV. Survival Odds to Minimize Risk Heterogeneity Bias in Heart Failure Trials: Application to Dapagliflozin. Circ Heart Fail. 2025 Dec;18(12):e013496. doi: 10.1161/CIRCHEARTFAILURE.125.013496. Epub 2025 Oct 31. PMID 41170566
- [Derived] McDowell K, Welsh P, Docherty KF, Morrow DA, Jhund PS, De Boer RA, O'Meara E, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Hammarstedt A, Langkilde AM, Solomon SD, Sattar N, Sabatine MS, McMurray JJV. Cellular Adhesion Molecules and Adverse Outcomes in Chronic Heart Failure: Findings From the DAPA-HF Randomized Clinical Trial. JAMA Cardiol. 2025 Aug 1;10(8):797-808. doi: 10.1001/jamacardio.2025.1592. PMID 40465275
- [Derived] Docherty KF, McDowell K, Welsh P, Petrie MC, Anand I, Berg DD, de Boer RA, Kober L, Kosiborod MN, Martinez FA, O'Meara E, Morrow DA, Ponikowski P, Sabatine MS, Sattar N, Schou M, Hammarstedt A, Sjostrand M, Langkilde AM, Jhund PS, Solomon SD, McMurray JJV. Interleukin-6 in Heart Failure With Reduced Ejection Fraction and the Effect of Dapagliflozin: An Exploratory Analysis of the Dapagliflozin and Prevention of Adverse Outcomes in Heart Failure Trial. JACC Heart Fail. 2025 Jul;13(7):102393. doi: 10.1016/j.jchf.2024.12.012. Epub 2025 Mar 12. PMID 40088234
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Kondo T, Mogensen UM, Talebi A, Gasparyan SB, Campbell RT, Docherty KF, de Boer RA, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Sabatine MS, Bengtsson O, Sjostrand M, Vaduganathan M, Solomon SD, Jhund PS, McMurray JJV. Dapagliflozin and Days of Full Health Lost in the DAPA-HF Trial. J Am Coll Cardiol. 2024 May 21;83(20):1973-1986. doi: 10.1016/j.jacc.2024.03.385. Epub 2024 Mar 25. PMID 38537918
- [Derived] Kondo T, Gasparyan SB, Jhund PS, Bengtsson O, Claggett BL, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Kober L, Lam CSP, Langkilde AM, Martinez FA, Petersson M, Ponikowski P, Sabatine MS, Shah SJ, Sjostrand M, Wilderang U, Vaduganathan M, Solomon SD, McMurray JJV. Use of Win Statistics to Analyze Outcomes in the DAPA-HF and DELIVER Trials. NEJM Evid. 2023 Nov;2(11):EVIDoa2300042. doi: 10.1056/EVIDoa2300042. Epub 2023 Oct 24. PMID 38320525
- [Derived] Kondo T, Butt JH, Curtain JP, Jhund PS, Docherty KF, Claggett BL, Vaduganathan M, Bachus E, Hernandez AF, Lam CSP, Inzucchi SE, Martinez FA, de Boer RA, Kosiborod MN, Desai AS, Kober L, Ponikowski P, Sabatine MS, Solomon SD, McMurray JJV. Efficacy of Dapagliflozin According to Heart Rate: A Patient-Level Pooled Analysis of DAPA-HF and DELIVER. Circ Heart Fail. 2023 Dec;16(12):e010898. doi: 10.1161/CIRCHEARTFAILURE.123.010898. Epub 2023 Oct 27. PMID 37886880
- [Derived] Docherty KF, McDowell K, Welsh P, Osmanska J, Anand I, de Boer RA, Kober L, Kosiborod MN, Martinez FA, O'Meara E, Ponikowski P, Schou M, Berg DD, Sabatine MS, Morrow DA, Jarolim P, Hammarstedt A, Sjostrand M, Langkilde AM, Solomon SD, Sattar N, Jhund PS, McMurray JJV. Association of Carbohydrate Antigen 125 on the Response to Dapagliflozin in Patients With Heart Failure. J Am Coll Cardiol. 2023 Jul 11;82(2):142-157. doi: 10.1016/j.jacc.2023.05.011. PMID 37407113
- [Derived] Butt JH, Docherty KF, Kosiborod MN, Inzucchi SE, Kober L, Langkilde AM, Martinez FA, Bengtsson O, Ponikowski P, Sabatine MS, Sjostrand M, Solomon S, Jhund PS, McMurray JJV. Dapagliflozin and Physical and Social Activity Limitations in Heart Failure With Reduced Ejection Fraction. JACC Heart Fail. 2023 Oct;11(10):1411-1423. doi: 10.1016/j.jchf.2023.04.016. Epub 2023 Jun 14. PMID 37318419
- [Derived] Butt JH, Kondo T, Yang M, Jhund PS, Docherty KF, Vaduganathan M, Claggett BL, Hernandez AF, Lam CSP, Inzucchi SE, Martinez FA, de Boer RA, Kosiborod MN, Desai AS, Kober L, Ponikowski P, Sabatine MS, Shah SJ, Zaozerska N, Wilderang U, Bengtsson O, Solomon SD, McMurray JJV. Heart failure, peripheral artery disease, and dapagliflozin: a patient-level meta-analysis of DAPA-HF and DELIVER. Eur Heart J. 2023 Jun 25;44(24):2170-2183. doi: 10.1093/eurheartj/ehad276. PMID 37220172
- [Derived] Bhatt AS, Kosiborod MN, Vaduganathan M, Claggett BL, Miao ZM, Kulac IJ, Lam CSP, Hernandez AF, Martinez F, Inzucchi SE, Shah SJ, de Boer RA, Jhund PS, Desai AS, Petersson M, Langkilde AM, McMurray JJV, Solomon SD. Effect of dapagliflozin on health status and quality of life across the spectrum of ejection fraction: Participant-level pooled analysis from the DAPA-HF and DELIVER trials. Eur J Heart Fail. 2023 Jul;25(7):981-988. doi: 10.1002/ejhf.2909. Epub 2023 Jun 7. PMID 37211977
- [Derived] Chatur S, Kondo T, Claggett BL, Docherty K, Miao ZM, Desai AS, Jhund PS, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez FA, Shah SJ, Petersson M, Langkilde AM, McMurray JJV, Solomon SD, Vaduganathan M. Effects of dapagliflozin on heart failure hospitalizations according to severity of inpatient course: Insights from DELIVER and DAPA-HF. Eur J Heart Fail. 2023 Aug;25(8):1364-1371. doi: 10.1002/ejhf.2912. Epub 2023 Jun 8. PMID 37210608
- [Derived] Yeoh SE, Docherty KF, Campbell RT, Jhund PS, Hammarstedt A, Heerspink HJL, Jarolim P, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Solomon SD, Sjostrand M, Bengtsson O, Greasley PJ, Sattar N, Welsh P, Sabatine MS, Morrow DA, McMurray JJV. Endothelin-1, Outcomes in Patients With Heart Failure and Reduced Ejection Fraction, and Effects of Dapagliflozin: Findings From DAPA-HF. Circulation. 2023 May 30;147(22):1670-1683. doi: 10.1161/CIRCULATIONAHA.122.063327. Epub 2023 Apr 11. PMID 37039015
- [Derived] Butt JH, Docherty KF, Claggett BL, Desai AS, Fang JC, Petersson M, Langkilde AM, de Boer RA, Cabrera Honorio JW, Hernandez AF, Inzucchi SE, Kosiborod MN, Kober L, Lam CSP, Martinez FA, Ponikowski P, Sabatine MS, Vardeny O, O'Meara E, Saraiva JFK, Shah SJ, Vaduganathan M, Jhund PS, Solomon SD, McMurray JJV. Dapagliflozin in Black and White Patients With Heart Failure Across the Ejection Fraction Spectrum. JACC Heart Fail. 2023 Apr;11(4):375-388. doi: 10.1016/j.jchf.2022.11.014. Epub 2023 Feb 1. PMID 36881399
- [Derived] Butt JH, Docherty KF, Claggett BL, Desai AS, Petersson M, Langkilde AM, de Boer RA, Hernandez AF, Inzucchi SE, Kosiborod MN, Kober L, Lam CSP, Martinez FA, Ponikowski P, Sabatine MS, Shah SJ, Vaduganathan M, Jhund PS, Solomon SD, McMurray JJV. Association of Dapagliflozin Use With Clinical Outcomes and the Introduction of Uric Acid-Lowering Therapy and Colchicine in Patients With Heart Failure With and Without Gout: A Patient-Level Pooled Meta-analysis of DAPA-HF and DELIVER. JAMA Cardiol. 2023 Apr 1;8(4):386-393. doi: 10.1001/jamacardio.2022.5608. PMID 36811901
- [Derived] Adamson C, Welsh P, Docherty KF, de Boer RA, Diez M, Drozdz J, Dukat A, Inzucchi SE, Kober L, Kosiborod MN, Ljungman CEA, Martinez FA, Ponikowski P, Sabatine MS, Morrow DA, Lindholm D, Hammarstedt A, Boulton DW, Greasley PJ, Langkilde AM, Solomon SD, Sattar N, McMurray JJV, Jhund PS. IGFBP-7 and Outcomes in Heart Failure With Reduced Ejection Fraction: Findings From DAPA-HF. JACC Heart Fail. 2023 Mar;11(3):291-304. doi: 10.1016/j.jchf.2022.09.004. Epub 2022 Nov 9. PMID 36592046
- [Derived] Docherty KF, Anand IS, Chiang CE, Chopra VK, Desai AS, Kitakaze M, Verma S, Vinh PN, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Bengtsson O, Ponikowski P, Sabatine MS, Sjostrand M, Solomon SD, Langkilde AM, Jhund PS, McMurray JJV. Effects of Dapagliflozin in Asian Patients With Heart Failure and Reduced Ejection Fraction in DAPA-HF. JACC Asia. 2022 Mar 29;2(2):139-153. doi: 10.1016/j.jacasi.2022.02.004. eCollection 2022 Apr. PMID 36339117
- [Derived] Desai AS, Jhund PS, Claggett BL, Vaduganathan M, Miao ZM, Kondo T, Barkoudah E, Brahimi A, Connolly E, Finn P, Lang NN, Mc Causland FR, McGrath M, Petrie MC, McMurray JJV, Solomon SD. Effect of Dapagliflozin on Cause-Specific Mortality in Patients With Heart Failure Across the Spectrum of Ejection Fraction: A Participant-Level Pooled Analysis of DAPA-HF and DELIVER. JAMA Cardiol. 2022 Dec 1;7(12):1227-1234. doi: 10.1001/jamacardio.2022.3736. PMID 36189985
- [Derived] Adamson C, Cowan LM, de Boer RA, Diez M, Drozdz J, Dukat A, Inzucchi SE, Kober L, Kosiborod MN, Ljungman CEA, Martinez FA, Ponikowski P, Sabatine MS, Lindholm D, Bengtsson O, Boulton DW, Greasley PJ, Langkilde AM, Sjostrand M, Solomon SD, McMurray JJV, Jhund PS. Liver tests and outcomes in heart failure with reduced ejection fraction: findings from DAPA-HF. Eur J Heart Fail. 2022 Oct;24(10):1856-1868. doi: 10.1002/ejhf.2649. Epub 2022 Aug 22. PMID 36054568
- [Derived] Docherty KF, Welsh P, Verma S, De Boer RA, O'Meara E, Bengtsson O, Kober L, Kosiborod MN, Hammarstedt A, Langkilde AM, Lindholm D, Little DJ, Sjostrand M, Martinez FA, Ponikowski P, Sabatine MS, Morrow DA, Schou M, Solomon SD, Sattar N, Jhund PS, McMurray JJV; DAPA-HF Investigators and Committees. Iron Deficiency in Heart Failure and Effect of Dapagliflozin: Findings From DAPA-HF. Circulation. 2022 Sep 27;146(13):980-994. doi: 10.1161/CIRCULATIONAHA.122.060511. Epub 2022 Aug 16. PMID 35971840
- [Derived] Butt JH, Dewan P, DeFilippis EM, Biering-Sorensen T, Docherty KF, Jhund PS, Kosiborod MN, Martinez FA, Bengtsson O, Johansen ND, Langkilde AM, Sjostrand M, Vaduganathan M, Solomon SD, Sabatine MS, Kober L, Fiuzat M, McMurray JJV. Effects of Dapagliflozin According to the Heart Failure Collaboratory Medical Therapy Score: Insights From DAPA-HF. JACC Heart Fail. 2022 Aug;10(8):543-555. doi: 10.1016/j.jchf.2022.03.009. Epub 2022 Jun 8. PMID 35902157
- [Derived] Yeoh SE, Docherty KF, Jhund PS, Petrie MC, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Bengtsson O, Boulton DW, Greasley PJ, Langkilde AM, Sjostrand M, Solomon SD, McMurray JJV. Relationship of Dapagliflozin With Serum Sodium: Findings From the DAPA-HF Trial. JACC Heart Fail. 2022 May;10(5):306-318. doi: 10.1016/j.jchf.2022.01.019. Epub 2022 Apr 6. PMID 35483792
- [Derived] Butt JH, Dewan P, Merkely B, Belohlavek J, Drozdz J, Kitakaze M, Inzucchi SE, Kosiborod MN, Martinez FA, Tereshchenko S, Ponikowski P, Bengtsson O, Lindholm D, Langkilde AM, Schou M, Sjostrand M, Solomon SD, Sabatine MS, Chiang CE, Docherty KF, Jhund PS, Kober L, McMurray JJV. Efficacy and Safety of Dapagliflozin According to Frailty in Heart Failure With Reduced Ejection Fraction : A Post Hoc Analysis of the DAPA-HF Trial. Ann Intern Med. 2022 Jun;175(6):820-830. doi: 10.7326/M21-4776. Epub 2022 Apr 26. PMID 35467935
- [Derived] Adamson C, Docherty KF, Heerspink HJL, de Boer RA, Damman K, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Petrie MC, Ponikowski P, Sabatine MS, Schou M, Solomon SD, Verma S, Bengtsson O, Langkilde AM, Sjostrand M, Vaduganathan M, Jhund PS, McMurray JJV. Initial Decline (Dip) in Estimated Glomerular Filtration Rate After Initiation of Dapagliflozin in Patients With Heart Failure and Reduced Ejection Fraction: Insights From DAPA-HF. Circulation. 2022 Aug 9;146(6):438-449. doi: 10.1161/CIRCULATIONAHA.121.058910. Epub 2022 Apr 20. PMID 35442064
- [Derived] Docherty KF, Simpson J, Jhund PS, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Bengtsson O, Sjostrand M, Lindholm D, Langkilde AM, Solomon SD, McMurray JJV; DAPA-HF Investigators and Committees. Effect of Dapagliflozin, Compared With Placebo, According to Baseline Risk in DAPA-HF. JACC Heart Fail. 2022 Feb;10(2):104-118. doi: 10.1016/j.jchf.2021.09.002. Epub 2022 Jan 12. PMID 35115084
- [Derived] Docherty KF, Ogunniyi MO, Anand IS, Desai AS, Diez M, Howlett JG, Nicolau JC, O'Meara E, Verma S, Inzucchi SE, Kober L, Kosiborod MN, Lindholm D, Martinez FA, Bengtsson O, Ponikowski P, Sabatine MS, Sjostrand M, Solomon SD, Langkilde AM, Jhund PS, McMurray JJV. Efficacy of Dapagliflozin in Black Versus White Patients With Heart Failure and Reduced Ejection Fraction. JACC Heart Fail. 2022 Jan;10(1):52-64. doi: 10.1016/j.jchf.2021.08.006. Epub 2021 Nov 10. PMID 34969498
- [Derived] Ryden L, Ferrannini G. Is the impact of add on heart failure therapy influenced by background therapy? Lancet Diabetes Endocrinol. 2022 Jan;10(1):3-5. doi: 10.1016/S2213-8587(21)00311-9. Epub 2021 Nov 30. No abstract available. PMID 34861151
- [Derived] Butt JH, Adamson C, Docherty KF, de Boer RA, Petrie MC, Inzucchi SE, Kosiborod MN, Maria Langkilde A, Lindholm D, Martinez FA, Bengtsson O, Schou M, O'Meara E, Ponikowski P, Sabatine MS, Sjostrand M, Solomon SD, Jhund PS, McMurray JJV, Kober L. Efficacy and Safety of Dapagliflozin in Heart Failure With Reduced Ejection Fraction According to N-Terminal Pro-B-Type Natriuretic Peptide: Insights From the DAPA-HF Trial. Circ Heart Fail. 2021 Dec;14(12):e008837. doi: 10.1161/CIRCHEARTFAILURE.121.008837. Epub 2021 Nov 22. PMID 34802253
- [Derived] Berg DD, Docherty KF, Sattar N, Jarolim P, Welsh P, Jhund PS, Anand IS, Chopra V, de Boer RA, Kosiborod MN, Nicolau JC, O'Meara E, Schou M, Hammarstedt A, Langkilde AM, Lindholm D, Sjostrand M, McMurray JJV, Sabatine MS, Morrow DA. Serial Assessment of High-Sensitivity Cardiac Troponin and the Effect of Dapagliflozin in Patients With Heart Failure With Reduced Ejection Fraction: An Analysis of the DAPA-HF Trial. Circulation. 2022 Jan 18;145(3):158-169. doi: 10.1161/CIRCULATIONAHA.121.057852. Epub 2021 Nov 8. PMID 34743554
- [Derived] Curtain JP, Docherty KF, Jhund PS, Petrie MC, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Bengtsson O, Langkilde AM, Sjostrand M, Solomon SD, McMurray JJV. Effect of dapagliflozin on ventricular arrhythmias, resuscitated cardiac arrest, or sudden death in DAPA-HF. Eur Heart J. 2021 Sep 21;42(36):3727-3738. doi: 10.1093/eurheartj/ehab560. PMID 34448003
- [Derived] Docherty KF, Jhund PS, Claggett B, Ferreira JP, Bengtsson O, Inzucchi SE, Kober L, Kosiborod MN, Langkilde AM, Martinez FA, Ponikowski P, Sabatine MS, Sjostrand M, Solomon SD, McMurray JJV; DAPA-HF Investigators and Committees. Extrapolating Long-term Event-Free and Overall Survival With Dapagliflozin in Patients With Heart Failure and Reduced Ejection Fraction: An Exploratory Analysis of a Phase 3 Randomized Clinical Trial. JAMA Cardiol. 2021 Nov 1;6(11):1298-1305. doi: 10.1001/jamacardio.2021.2632. PMID 34319398
- [Derived] Adamson C, Jhund PS, Docherty KF, Belohlavek J, Chiang CE, Diez M, Drozdz J, Dukat A, Howlett J, Ljungman CEA, Petrie MC, Schou M, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Solomon SD, Bengtsson O, Langkilde AM, Lindholm D, Sjostrand M, McMurray JJV. Efficacy of dapagliflozin in heart failure with reduced ejection fraction according to body mass index. Eur J Heart Fail. 2021 Oct;23(10):1662-1672. doi: 10.1002/ejhf.2308. Epub 2021 Jul 29. PMID 34272791
- [Derived] Jhund PS, Ponikowski P, Docherty KF, Gasparyan SB, Bohm M, Chiang CE, Desai AS, Howlett J, Kitakaze M, Petrie MC, Verma S, Bengtsson O, Langkilde AM, Sjostrand M, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Sabatine MS, Solomon SD, McMurray JJV. Dapagliflozin and Recurrent Heart Failure Hospitalizations in Heart Failure With Reduced Ejection Fraction: An Analysis of DAPA-HF. Circulation. 2021 May 18;143(20):1962-1972. doi: 10.1161/CIRCULATIONAHA.121.053659. Epub 2021 Apr 9. PMID 33832352
- [Derived] Butt JH, Docherty KF, Petrie MC, Schou M, Kosiborod MN, O'Meara E, Katova T, Ljungman CEA, Diez M, Ogunniyi MO, Langkilde AM, Sjostrand M, Lindholm D, Bengtsson O, Martinez FA, Ponikowski P, Sabatine MS, Solomon SD, Jhund PS, McMurray JJV, Kober L. Efficacy and Safety of Dapagliflozin in Men and Women With Heart Failure With Reduced Ejection Fraction: A Prespecified Analysis of the Dapagliflozin and Prevention of Adverse Outcomes in Heart Failure Trial. JAMA Cardiol. 2021 Jun 1;6(6):678-689. doi: 10.1001/jamacardio.2021.0379. PMID 33787831
- [Derived] Berg DD, Jhund PS, Docherty KF, Murphy SA, Verma S, Inzucchi SE, Kober L, Kosiborod MN, Langkilde AM, Martinez FA, Bengtsson O, Ponikowski P, Sjostrand M, Solomon SD, McMurray JJV, Sabatine MS. Time to Clinical Benefit of Dapagliflozin and Significance of Prior Heart Failure Hospitalization in Patients With Heart Failure With Reduced Ejection Fraction. JAMA Cardiol. 2021 May 1;6(5):499-507. doi: 10.1001/jamacardio.2020.7585. PMID 33595593
- [Derived] Shen L, Kristensen SL, Bengtsson O, Bohm M, de Boer RA, Docherty KF, Inzucchi SE, Katova T, Kober L, Kosiborod MN, Langkilde AM, Lindholm D, Martinez MFA, O'Meara E, Nicolau JC, Petrie MC, Ponikowski P, Sabatine MS, Schou M, Sjostrand M, Solomon SD, Jhund PS, McMurray JJV. Dapagliflozin in HFrEF Patients Treated With Mineralocorticoid Receptor Antagonists: An Analysis of DAPA-HF. JACC Heart Fail. 2021 Apr;9(4):254-264. doi: 10.1016/j.jchf.2020.11.009. Epub 2021 Feb 3. PMID 33549554
- [Derived] Dewan P, Docherty KF, Bengtsson O, de Boer RA, Desai AS, Drozdz J, Hawkins NM, Inzucchi SE, Kitakaze M, Kober L, Kosiborod MN, Langkilde AM, Lindholm D, Martinez FA, Merkely B, Petrie MC, Ponikowski P, Sabatine MS, Schou M, Sjostrand M, Solomon SD, Verma S, Jhund PS, McMurray JJV. Effects of dapagliflozin in heart failure with reduced ejection fraction and chronic obstructive pulmonary disease: an analysis of DAPA-HF. Eur J Heart Fail. 2021 Apr;23(4):632-643. doi: 10.1002/ejhf.2083. Epub 2021 Jan 18. PMID 33368858
- [Derived] Inzucchi SE, Docherty KF, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Solomon SD, Verma S, Belohlavek J, Bohm M, Chiang CE, de Boer RA, Diez M, Dukat A, Ljungman CEA, Bengtsson O, Langkilde AM, Sjostrand M, Jhund PS, McMurray JJV; DAPA-HF Investigators and Committees. Dapagliflozin and the Incidence of Type 2 Diabetes in Patients With Heart Failure and Reduced Ejection Fraction: An Exploratory Analysis From DAPA-HF. Diabetes Care. 2021 Feb;44(2):586-594. doi: 10.2337/dc20-1675. Epub 2020 Dec 18. PMID 33355302
- [Derived] Yeoh SE, Dewan P, Jhund PS, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Solomon SD, Bengtsson O, Sjostrand M, Langkilde AM, McMurray JJV; DAPA-HF Investigators and Committees. Patient Characteristics, Clinical Outcomes, and Effect of Dapagliflozin in Relation to Duration of Heart Failure: Is It Ever Too Late to Start a New Therapy? Circ Heart Fail. 2020 Dec;13(12):e007879. doi: 10.1161/CIRCHEARTFAILURE.120.007879. Epub 2020 Nov 9. PMID 33164553
- [Derived] Docherty KF, Jhund PS, Bengtsson O, DeMets DL, Inzucchi SE, Kober L, Kosiborod MN, Langkilde AM, Martinez FA, Sabatine MS, Sjostrand M, Solomon SD, McMurray JJV; DAPA-HF Investigators and Committees. Effect of Dapagliflozin in DAPA-HF According to Background Glucose-Lowering Therapy. Diabetes Care. 2020 Nov;43(11):2878-2881. doi: 10.2337/dc20-1402. Epub 2020 Sep 2. PMID 33082245
- [Derived] Jhund PS, Solomon SD, Docherty KF, Heerspink HJL, Anand IS, Bohm M, Chopra V, de Boer RA, Desai AS, Ge J, Kitakaze M, Merkley B, O'Meara E, Shou M, Tereshchenko S, Verma S, Vinh PN, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Bengtsson O, Langkilde AM, Sjostrand M, McMurray JJV. Efficacy of Dapagliflozin on Renal Function and Outcomes in Patients With Heart Failure With Reduced Ejection Fraction: Results of DAPA-HF. Circulation. 2021 Jan 26;143(4):298-309. doi: 10.1161/CIRCULATIONAHA.120.050391. Epub 2020 Oct 12. PMID 33040613
- [Derived] Docherty KF, Jhund PS, Anand I, Bengtsson O, Bohm M, de Boer RA, DeMets DL, Desai AS, Drozdz J, Howlett J, Inzucchi SE, Johanson P, Katova T, Kober L, Kosiborod MN, Langkilde AM, Lindholm D, Martinez FA, Merkely B, Nicolau JC, O'Meara E, Ponikowski P, Sabatine MS, Sjostrand M, Solomon SD, Tereshchenko S, Verma S, McMurray JJV. Effect of Dapagliflozin on Outpatient Worsening of Patients With Heart Failure and Reduced Ejection Fraction: A Prespecified Analysis of DAPA-HF. Circulation. 2020 Oct 27;142(17):1623-1632. doi: 10.1161/CIRCULATIONAHA.120.047480. Epub 2020 Sep 4. PMID 32883108
- [Derived] Serenelli M, Bohm M, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Solomon SD, DeMets DL, Bengtsson O, Sjostrand M, Langkilde AM, Anand IS, Chiang CE, Chopra VK, de Boer RA, Diez M, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Verma S, Docherty KF, Jhund PS, McMurray JJV. Effect of dapagliflozin according to baseline systolic blood pressure in the Dapagliflozin and Prevention of Adverse Outcomes in Heart Failure trial (DAPA-HF). Eur Heart J. 2020 Sep 21;41(36):3402-3418. doi: 10.1093/eurheartj/ehaa496. PMID 32820334
- [Derived] Jackson AM, Dewan P, Anand IS, Belohlavek J, Bengtsson O, de Boer RA, Bohm M, Boulton DW, Chopra VK, DeMets DL, Docherty KF, Dukat A, Greasley PJ, Howlett JG, Inzucchi SE, Katova T, Kober L, Kosiborod MN, Langkilde AM, Lindholm D, Ljungman CEA, Martinez FA, O'Meara E, Sabatine MS, Sjostrand M, Solomon SD, Tereshchenko S, Verma S, Jhund PS, McMurray JJV. Dapagliflozin and Diuretic Use in Patients With Heart Failure and Reduced Ejection Fraction in DAPA-HF. Circulation. 2020 Sep 15;142(11):1040-1054. doi: 10.1161/CIRCULATIONAHA.120.047077. Epub 2020 Jul 16. PMID 32673497
- [Derived] Solomon SD, Jhund PS, Claggett BL, Dewan P, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Inzucchi SE, Desai AS, Bengtsson O, Lindholm D, Sjostrand M, Langkilde AM, McMurray JJV. Effect of Dapagliflozin in Patients With HFrEF Treated With Sacubitril/Valsartan: The DAPA-HF Trial. JACC Heart Fail. 2020 Oct;8(10):811-818. doi: 10.1016/j.jchf.2020.04.008. Epub 2020 Jul 8. PMID 32653447
- [Derived] Dewan P, Solomon SD, Jhund PS, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, DeMets DL, Sabatine MS, Bengtsson O, Sjostrand M, Langkilde AM, Anand IS, Belohlavek J, Chopra VK, Dukat A, Kitakaze M, Merkely B, O'Meara E, Schou M, Vinh PN, McMurray JJV; DAPA-HF Investigators and Committees. Efficacy and safety of sodium-glucose co-transporter 2 inhibition according to left ventricular ejection fraction in DAPA-HF. Eur J Heart Fail. 2020 Jul;22(7):1247-1258. doi: 10.1002/ejhf.1867. Epub 2020 Jun 15. PMID 32539224
- [Derived] Petrie MC, Verma S, Docherty KF, Inzucchi SE, Anand I, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett J, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Vinh PN, Schou M, Tereshchenko S, Kober L, Kosiborod MN, Langkilde AM, Martinez FA, Ponikowski P, Sabatine MS, Sjostrand M, Solomon SD, Johanson P, Greasley PJ, Boulton D, Bengtsson O, Jhund PS, McMurray JJV. Effect of Dapagliflozin on Worsening Heart Failure and Cardiovascular Death in Patients With Heart Failure With and Without Diabetes. JAMA. 2020 Apr 14;323(14):1353-1368. doi: 10.1001/jama.2020.1906. PMID 32219386
- [Derived] Kosiborod MN, Jhund PS, Docherty KF, Diez M, Petrie MC, Verma S, Nicolau JC, Merkely B, Kitakaze M, DeMets DL, Inzucchi SE, Kober L, Martinez FA, Ponikowski P, Sabatine MS, Solomon SD, Bengtsson O, Lindholm D, Niklasson A, Sjostrand M, Langkilde AM, McMurray JJV. Effects of Dapagliflozin on Symptoms, Function, and Quality of Life in Patients With Heart Failure and Reduced Ejection Fraction: Results From the DAPA-HF Trial. Circulation. 2020 Jan 14;141(2):90-99. doi: 10.1161/CIRCULATIONAHA.119.044138. Epub 2019 Nov 17. PMID 31736335
- [Derived] Martinez FA, Serenelli M, Nicolau JC, Petrie MC, Chiang CE, Tereshchenko S, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Ponikowski P, Sabatine MS, DeMets DL, Dutkiewicz-Piasecka M, Bengtsson O, Sjostrand M, Langkilde AM, Jhund PS, McMurray JJV. Efficacy and Safety of Dapagliflozin in Heart Failure With Reduced Ejection Fraction According to Age: Insights From DAPA-HF. Circulation. 2020 Jan 14;141(2):100-111. doi: 10.1161/CIRCULATIONAHA.119.044133. Epub 2019 Nov 17. PMID 31736328
- [Derived] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Derived] McMurray JJV, DeMets DL, Inzucchi SE, Kober L, Kosiborod MN, Langkilde AM, Martinez FA, Bengtsson O, Ponikowski P, Sabatine MS, Sjostrand M, Solomon SD; DAPA-HF Committees and Investigators. The Dapagliflozin And Prevention of Adverse-outcomes in Heart Failure (DAPA-HF) trial: baseline characteristics. Eur J Heart Fail. 2019 Nov;21(11):1402-1411. doi: 10.1002/ejhf.1548. Epub 2019 Jul 15. PMID 31309699
- [Derived] Nassif ME, Kosiborod M. Effects of sodium glucose cotransporter type 2 inhibitors on heart failure. Diabetes Obes Metab. 2019 Apr;21 Suppl 2:19-23. doi: 10.1111/dom.13678. PMID 31081589
- See also: redacted protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1699C00001&attachmentIdentifier=66b47cad-8320-450c-8663-8298a1e7f535&fileName=D1699C00001_Protocol_redacted.pdf&versionIdentifier=
- See also: redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1699C00001&attachmentIdentifier=0dea388e-44d4-4c23-9555-8aea2ea3448d&fileName=D1699C00001_Statistical_Analysis_Plan_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapa 10mg: Dapagliflozin 10 mg, given once daily per oral use.
- Placebo: Placebo tablet to match dapagliflozin 10 mg, given once daily per oral use.
Period: Overall Study
Arm/Group | Dapa 10mg | Placebo
Started | 2373 | 2371
Completed | 2368 | 2365
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapa 10mg | Placebo | Total
Number analyzed (Participants) | 2373 | 2371 | 4744
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (11.0) | 66.5 (10.8) | 66.3 (10.9)
Age, Customized [Count of Participants; unit: Participants]
  <=50 | 208 | 188 | 396
  >50 | 2165 | 2183 | 4348
Age, Customized [Count of Participants; unit: Participants]
  <=65 | 1032 | 998 | 2030
  >65 | 1341 | 1373 | 2714
Age, Customized [Count of Participants; unit: Participants]
  <=65 | 1032 | 998 | 2030
  66 - 75 | 825 | 886 | 1711
  >75 | 516 | 487 | 1003
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 564 | 545 | 1109
  Male | 1809 | 1826 | 3635
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 381 | 387 | 768
  Not Hispanic or Latino | 1992 | 1984 | 3976
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1662 | 1671 | 3333
  Black or African American | 122 | 104 | 226
  Asian | 552 | 564 | 1116
  Native Hawaiian or other Pacific Islander | 0 | 2 | 2
  American Indian or Alaska Native | 3 | 1 | 4
  Other | 34 | 29 | 63
Main etiology of HF [Count of Participants; unit: Participants]
  Ischaemic | 1316 | 1358 | 2674
  Non-Ischaemic | 857 | 830 | 1687
  Unknown | 200 | 183 | 383
Prior HF hospitalization [Count of Participants; unit: Participants]
  Yes | 1124 | 1127 | 2251
NYHA class at enrollment [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Functional Classification places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina. A higher class means a worse functional condition.
  Participants
    II | 1606 | 1597 | 3203
    III | 747 | 751 | 1498
    IV | 20 | 23 | 43
Type 2 diabetes at baseline [Count of Participants; unit: Participants]
  Yes | 1075 | 1064 | 2139
  No | 1298 | 1307 | 2605
LVEF [Mean (Standard Deviation); unit: Percentage of blood leaving the heart] | 31.2 (6.7) | 30.9 (6.9) | 31.1 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Subjects Included in the Composite Endpoint of CV Death, Hospitalization Due to Heart Failure or Urgent Visit Due to Heart Failure.
Description: Primary efficacy
Time Frame: Up to 27.8 months.
Measure: Count of Participants; unit: Participants
Groups:
- Dapa 10 mg: Dapagliflozin 10 mg tablets administered orally once daily
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 2373 | 2371
Participants | 386 | 502
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Regression, Cox; Stratified by Type 2 Diabetes status at randomization and including the history of hospitalizations due to Heart failure as a factor; Hazard Ratio (HR) = 0.74, 95% CI [0.65 to 0.85]

2. Secondary Outcome: Subjects Included in the Composite Endpoint of CV Death or Hospitalization Due to Heart Failure.
Description: Secondary
Time Frame: Up to 27.8 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 2373 | 2371
Participants | 382 | 495
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.75, 95% CI [0.65 to 0.85]

3. Secondary Outcome: Events Included in the Composite Endpoint of Recurrent Hospitalizations Due to Heart Failure and CV Death.
Description: Secondary
Time Frame: Up to 27.8 months.
Measure: Number; unit: events
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 2373 | 2371
events | 567 | 742
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.0002, LWYY proportional rates model; [statistical method as in outcome 1, analysis 1]; Rate Ratio (RR) = 0.75, 95% CI [0.65 to 0.88]

4. Secondary Outcome: Change From Baseline in the KCCQ Total Symptom Score
Description: KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The KCCQ total symptom score incorporates the symptom domains into a single score. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline and 8 months or death before 8 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 2373 | 2371
Scores on a scale | 6.1 (18.6) | 3.3 (19.2)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Win Ratio — The p-value is obtained from a rank ANCOVA adjusted for baseline KCCQ score and stratified by T2DM status at randomization; Stratified by Type 2 Diabetes status at randomization and including baseline score as a covariate; Win Ratio (WR) = 1.18, 95% CI [1.11 to 1.26] — The composite of change from baseline in total symptom score at 8 months, or death before 8 months

5. Secondary Outcome: Subjects Included in the Composite Endpoint of ≥50% Sustained Decline in eGFR, ESRD or Renal Death.
Description: Secondary
Time Frame: Up to 27.8 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 2373 | 2371
Participants | 28 | 39
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.1681, Regression, Cox; Stratified by Type 2 Diabetes status at randomization and including baseline eGFR as a covariate; Hazard Ratio (HR) = 0.71, 95% CI [0.44 to 1.16]

6. Secondary Outcome: Subjects Included in the Endpoint of All-cause Mortality.
Description: Secondary
Time Frame: Up to 27.8 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapa 10 mg | Placebo
Number analyzed (Participants) | 2373 | 2371
Participants | 276 | 329
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.0217, Regression, Cox; Stratified by Type 2 Diabetes status at randomization; Hazard Ratio (HR) = 0.83, 95% CI [0.71 to 0.97]

ADVERSE EVENTS:
Time Frame: Up to 28.3 months.
Description: For analysis of Adverse Events Safety analysis set is used. Safety analysis set : Consisted of all randomized patients who received at least one dose of study drug.
Arm/Group | Dapa 10mg | Placebo
All-Cause Mortality (participants affected / at risk) | 286/2368 | 333/2368
Serious Adverse Events (participants affected / at risk) | 895/2368 | 994/2368
Other Adverse Events (participants affected / at risk) | 299/2368 | 325/2368
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapa 10mg (N=2368) | Placebo (N=2368)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 11 (13)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 5 (6) | 3 (3)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 37 (37) | 38 (40)
Angina pectoris (Cardiac disorders) | 12 (12) | 12 (12)
Angina unstable (Cardiac disorders) | 21 (24) | 30 (31)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 8 (8)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 26 (27) | 39 (43)
Atrial flutter (Cardiac disorders) | 8 (9) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 4 (4)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 7 (7)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 9 (9) | 10 (10)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 262 (380) | 351 (523)
Cardiac failure acute (Cardiac disorders) | 42 (58) | 59 (75)
Cardiac failure chronic (Cardiac disorders) | 27 (32) | 33 (46)
Cardiac failure congestive (Cardiac disorders) | 65 (102) | 70 (106)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 9 (10) | 15 (16)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 3 (3)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 4 (4)
Coronary artery disease (Cardiac disorders) | 9 (10) | 8 (8)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 3 (3)
Extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Frederick's syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 2 (2) | 4 (5)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 3 (3)
Myocardial fibrosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 16 (16) | 17 (17)
Myocardial ischaemia (Cardiac disorders) | 3 (3) | 4 (4)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 0 (0) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 3 (3)
Sinus node dysfunction (Cardiac disorders) | 3 (3) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 3 (3)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Torsade de pointes (Cardiac disorders) | 2 (2) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 6 (6) | 7 (8)
Ventricular extrasystoles (Cardiac disorders) | 4 (4) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 11 (11) | 6 (7)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 34 (41) | 54 (65)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 4 (4) | 8 (8)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (2)
Glaucoma (Eye disorders) | 1 (1) | 3 (3)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Strabismus (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 3 (4)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 5 (5)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (5) | 7 (7)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 9 (9) | 5 (5)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 6 (6) | 4 (4)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Asthenia (General disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 4 (4) | 5 (5)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 48 (48) | 48 (48)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Implant site haemorrhage (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Medical device site inflammation (General disorders) | 0 (0) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1)
Necrosis (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 6 (6) | 16 (19)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 18 (18) | 27 (27)
Sudden death (General disorders) | 19 (19) | 10 (10)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (2)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 4 (4)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 5 (5)
Cholecystitis acute (Hepatobiliary disorders) | 6 (6) | 8 (8)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 (3) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder enlargement (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Heart transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 2 (2)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 12 (13) | 6 (6)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cardiac infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 9 (11) | 10 (12)
Cellulitis gangrenous (Infections and infestations) | 1 (1) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 3 (3) | 3 (3)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2)
Endocarditis (Infections and infestations) | 1 (1) | 4 (4)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Endotoxic shock (Infections and infestations) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 3 (3)
Erysipelas (Infections and infestations) | 1 (2) | 4 (4)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 2 (5) | 6 (7)
Gastroenteritis (Infections and infestations) | 3 (3) | 6 (6)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Hiv infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (2) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 2 (2)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (3)
Intestinal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 4 (7) | 4 (4)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Mediastinal abscess (Infections and infestations) | 1 (1) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 7 (9) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Perichondritis (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 2 (2)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 76 (83) | 82 (87)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Pyelocystitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 1 (2)
Renal cyst infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 5 (5)
Rickettsiosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 13 (13) | 14 (14)
Septic shock (Infections and infestations) | 8 (9) | 8 (9)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 1 (2) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 3 (3) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (13) | 17 (17)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 4 (4) | 7 (7)
Wound infection (Infections and infestations) | 5 (5) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac valve rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 7 (7) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 4 (4) | 3 (3)
Blood glucose increased (Investigations) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 2 (2)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Pulmonary arterial pressure increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 2 (2) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 10 (10) | 8 (8)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (6) | 4 (4)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Diabetic ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 7 (7)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pleural mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 3 (3) | 2 (2)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 8 (9) | 11 (12)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 7 (7) | 5 (5)
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Embolic stroke (Nervous system disorders) | 1 (1) | 3 (3)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 3 (3) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Iiird nerve paresis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 24 (26) | 26 (28)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (2)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 3 (3)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 7 (7) | 13 (14)
Transient ischaemic attack (Nervous system disorders) | 13 (13) | 7 (7)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Vertebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (2) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device failure (Product Issues) | 0 (0) | 2 (2)
Device inappropriate shock delivery (Product Issues) | 0 (0) | 1 (1)
Device lead issue (Product Issues) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 2 (2)
Lead dislodgement (Product Issues) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar i disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 2 (2)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 23 (25) | 46 (49)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 0 (0) | 2 (3)
Chronic kidney disease (Renal and urinary disorders) | 4 (4) | 8 (10)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 8 (8) | 8 (9)
Renal impairment (Renal and urinary disorders) | 7 (7) | 13 (14)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 (5) | 2 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Orchitis noninfective (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 14 (16)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 22 (34)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal lesion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 14 (14)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (5)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary vasculitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0)
Angiodysplasia (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 2 (2) | 2 (2)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 2 (2)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 3 (3)
Circulatory collapse (Vascular disorders) | 1 (1) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 6 (7)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (2) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Haematocoele (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Hypertensive crisis (Vascular disorders) | 3 (3) | 3 (3)
Hypertensive emergency (Vascular disorders) | 0 (0) | 2 (2)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 7 (9) | 11 (12)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 5 (6)
Peripheral arterial occlusive disease (Vascular disorders) | 11 (11) | 10 (11)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 9 (11) | 5 (8)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapa 10mg (N=2368) | Placebo (N=2368)
Atrial fibrillation (Cardiac disorders) | 58 (63) | 52 (55)
Cardiac failure (Cardiac disorders) | 76 (90) | 130 (154)
Nasopharyngitis (Infections and infestations) | 63 (84) | 76 (100)
Renal impairment (Renal and urinary disorders) | 63 (67) | 56 (60)
Hypotension (Vascular disorders) | 88 (98) | 73 (81)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT03036124/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT03036124/SAP_001.pdf